CLINICAL TRIAL: NCT01352364
Title: Analysis Of Equilibrium And Motor Coordination Of Deaf Children's Pre And Post Intervention Physiotherapeutic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Sinos Valley (Other)
Responsible Party: Klaus Loges, Universidade do Vale do Rio dos Sinos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I01
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2009-07

CONDITIONS: Motor Skills in Deaf Children; Deafness
Keywords: Physiotherapy.; Deafness.; Postural balance.; Motor skills.
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- deaf children (Experimental)
  Interventions: Other: physiotherapy intervention

INTERVENTIONS:
Other: physiotherapy intervention — a program of physical therapy intervention can match or improve motor skills in the deaf children

SUMMARY:
This study aimed to assess and reassess the balance and motor skills of deaf children, passed six weeks of intervention and to verify whether a program of physical therapy intervention can match or improve motor skills. This study was quasi-experimental before and after, with 10 children from a school in Caxias do Sul / RS. Motor skills were evaluated using pre and post test KTK Coordination Body, and the activities were held once a week for six weeks in sessions of forty minutes. It was used for statistical analysis the Student t test dependent and independent (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* age 7 to 10 years of age.
* hearing disorders proven by presenting specific examination of Auditory Evoked Potential and Examination of the brainstem (Brainstem Evoked Response - Bera).
* consent of parents / guardians of children to participate in the study by signing Term of Informed Consent (IC).

Exclusion Criteria:

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Balance | two months

SECONDARY OUTCOMES:
motor coordination | two months

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Rombaldi Bernardi, Physiotherapist, Principal Investigator — University of the Sinos Valley
Locations (1):
- Municipal School For Elementary School Helen Keller, Caxias do Sul, Rio Grande do Sul, Brazil